CLINICAL TRIAL: NCT02239432
Title: Prospective Cohort Study of Telomere Biology Among Patients With Early Adenocarcinoma of the Lung
Brief Title: Telomere Biology in Early Adenocarcinoma of the Lung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0067-14-MMC
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Adenocarcinoma of the Lung; Adenocarcinoma, Bronchiolo-Alveolar
Keywords: Adenocarcinoma of the Lung; Adenocarcinoma, Bronchiolo-Alveolar
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One peripheral blood sample is taken for lymphocyte culture and subsequently telomere length and activity analysis (previously described, Laish I, Gene 2013;529:245-9)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Suspected Adenocarcinoma of the Lung: Patients with suspected adenocarcinoma of the lung referred for surgical lung biopsy after multi-disciplinary team recommendation.
- Healthy Control: Age and sex-matched patients with no known lung disease or other chronic inflammatory disease or malignancy
- Age-matched controls with proven solid lung malignancy: Patients with biopsy-proven advanced solid malignancy of the lung

SUMMARY:
Early adenocarcinoma of the lung has an excellent five-year survival after resection. However, its clinical and radiologic presentation is highly variable. Traditional means for preoperative diagnosis such as Positron Emission Tomography (PET-CT) and trans-thoracic needle biopsy demonstrate unacceptable false positive and negative rates.

Telomere biology is activated aberrantly is most lung cancers but has not been studied in early stages to the best of our knowledge.

The objective of this study is to evaluate telomere length and activity with suspected early stage adenocarcinoma of the lung.

DETAILED DESCRIPTION:
Bronchoalveolar carcinoma has been traditionally used to refer to a subset of adenocarcinoma distinguished by its peripheral location, typical "lepidic" growth pattern and tendency for both bronchogenic and lymphatic spread. For the purpose of this discussion and consistency with the revised 2011 criteria, BAC subtypes will be collectively referred to as early adenocarcinoma.

The clinical presentation of early adenocarcinoma subtypes is highly variable ranging from a small solitary nodule to extensive lobar consolidation. Many peripheral lesions have a characteristic ground glass opacity appearance on Chest CT, which may correlate with an improved prognosis. The reported five-year disease-free survival after resection for isolated lesions may approaches 100%.

Preoperative diagnosis of such lesions is complicated by several limitations. First, the differential diagnosis is broad including an extensive number of inflammatory and infectious processes. Second, positron emission tomography (PET), which identifies regions of increased metabolic activity, may be falsely negative due to the slow growth of early adenocarcinoma lesions. Transbronchial needle biopsy is also unreliable to confirm or exclude disease in non-solid type lesions.

The proportion of lung cancers classified as adenocarcinoma has steadily increased and now comprises nearly ½ of cases. However, the proportion of adenocarcinoma in situ is uncertain. Previous reports range from 5-10% in a large series to as high as 24% in the large Surveillance, Epidemiology and End Results database. Thus, these early adenocarcinoma lesions may represent a disproportionately large number of lung cancers which are PET negative yet carry an excellent prognosis after early resection. The early adenocarcinoma subtypes represent a clinical entity requiring further characterization to distinguish lesions more likely to be malignant from benign.

Telomerase is activated aberrantly in most lung cancers and mutations in telomerase components predispose to solid malignancies. For patients with non-small cell lung cancer, numerous studies correlate increased tumor telomerase activity with increased likelihood of Stage IIIB and Stage IV disease and/or reduced survival. Furthermore, telomerase inhibition is currently being studied in clinical trials of patients with advanced non-small lung cancer.

Problem:

The semi-solid lung lesion may represent early stage adenocarcinoma which has an excellent prognosis upon early diagnosis and prompt surgical resection. However, the semi-solid lesion has a broad differential diagnosis and preoperative features characteristic of adenocarcinoma are needed to distinguish malignant from benign lesions.

Objective:

To study telomere length and telomerase activity in patients with suspected early adenocarcinoma of the lung whom are referred for surgical biopsy of lung lesions.

ELIGIBILITY:
Inclusion Criteria:

Patients referred by a multi-disciplinary team meeting recommendation for surgical lung biopsy due to suspected adenocarcinoma of the lung and agree to a one-time peripheral blood sample for telomere analysis as described.

Exclusion Criteria:

Patients whom were not evaluated by the multi-disciplinary team discussion prior to referral for surgical lung biopsy.

Patients with other chronic inflammatory disease requiring immunosuppressive therapy or known extra-pulmonary malignancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred by a multi-disciplinary team meeting recommendation for surgical lung biopsy due to suspected adenocarcinoma of the lung.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Telomere Capture Percentage | one-time peripheral blood sample
  According to our previous experience with telomore biology in different disease states, we estimate a standard deviation (SD) of 1.3 of telomere capture (%) for the controls (healthy patients without known lung disease) and a SD of 2.4 (TC%) for biopsy-proven adenocarcinoma of the lung. For a clinically significance of at least 2%, we estimate a sample size of at least 16 patients with biopsy-proven disease to detect a statistically significant of 5% with a power of 80% (calculated by the independent t-test).

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Soroka University Medical Center, Beersheba
  - Meir Medical Center, Kfar Saba